CLINICAL TRIAL: NCT01840423
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Effects of Single and Repeated Escalating Doses of ODM-104: a Randomised, Double-blind, Placebo- and Entacapone-controlled Single Centre First-in-man Study in Healthy Volunteers.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ODM-104 in Healthy Volunteers
Acronym: NOCIFIM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 3112001
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: First in man study; Volunteer study
MeSH Terms: interventions — entacapone; carbidopa, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ODM-104 (Experimental): Oral capsules dosage 10-800mg once daily for one day or three times daily for 7 days
  Interventions: Drug: ODM-104
- Placebo (Placebo Comparator): Oral capsules given once daily for one day or three times daily for 7 days
  Interventions: Drug: Placebo
- entacapone + levodopa/carbidopa (Active Comparator): entacapone: oral tablet 200mg given four times daily for one day; levodopa/carbidopa: oral tablet 100/25mg given four times daily for one day
  Interventions: Drug: Entacapone; Drug: levodopa/carbidopa

INTERVENTIONS:
Drug: ODM-104 — ODM-104
  Arms: ODM-104
Drug: Placebo — Placebo
  Arms: Placebo
Drug: Entacapone — entacapone + levodopa/carbidopa
  Arms: entacapone + levodopa/carbidopa
Drug: levodopa/carbidopa — entacapone + levodopa/carbidopa
  Arms: entacapone + levodopa/carbidopa

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of escalating doses of ODM-104 when given to healthy male volunteers.

DETAILED DESCRIPTION:
The study is divided into two parts. Part one is a crossover study where healthy volunteers will receive two doses of ODM-104 and one dose of placebo. Part II of the study is a multiple ascending dose parallel group study where healthy volunteers will receive ODM-104 three times daily for seven days. Healthy volunteers taking part in Part II of the study will also receive levo/carbidopa and entacapone four times daily on day 1 and levo/carbidopa in addition to ODM-104 on day 9. The study will also look at the pharmacokinetic(how the body handles the drug) and pharmacodynamics (how the drug affects the body) of ODM-104.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects aged between 18 and 45 years
* BMI 18-30 kg/m2
* Weight 55-95kg
* Written informed consent
* Good General Health

Exclusion Criteria:

* Vulnerable subjects
* Veins unsuitable for repeated venipuncture
* Evidence of clinically significant cardiovascular, renal, hepatic, hematological, Gi, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disorder
* History of or positive test for drug abuse
* Any condition requiring regular concomitant medication
* Blood donation or significant loss of blood within 2 months prior to screening
* Abnormal 12 lead ECG finding of clinical relevance
* Heart rate (HR) <50bpm or >90bpm after 10 minutes in a supine position
* Systolic blood pressure <90mmHg or >140mmHg after 10 minutes in a supine position
* Diastolic blood pressure <50mmHg or >90mmHg after 10 minutes in a supine position
* Abnormal 24 hour Holter recording of clinical relevance at screening
* Any abnormal laboratory value, vital signs or physical examination causing a health risk to the volunteer

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Erythrocyte Catechol-O-methyltransferase (COMT) inhibition. | 0, 0.16, 0.33, 0.5, 0.75,1.0,1.5, 2, 3, 4, 6, 10, 16, 24h post dose
  Maximal COMT inhibition and area under the COMT inhibition curve (AUCC)

SECONDARY OUTCOMES:
Area under the plasma concentration curve (AUC) | 0, 0.16, 0.33, 0.5, 0.75, 1, 1.5, 2, 2, 4, 6, 10, 16, 24h post dose
  AUC under the plasma concentration curve

CONTACTS AND LOCATIONS:
Overall Officials: Rainard Fuhr, MD, Principal Investigator — Parexel; angela ruck, PhD, Study Director — Orion Corporation, Orion Pharma
Locations (1):
- Parexel International GmbH, Berlin, Germany